CLINICAL TRIAL: NCT07222813
Title: Performance of Liver Stiffness Measurement (LSM) by FibroScan® for the Diagnosis of Elevated Central Venous Pressure (CVP)
Brief Title: Evaluation of Liver Stiffness Performance, by FibroScan®, to Detect Elevated Central Venous Pressure (CVP)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cs002
Record Dates: First submitted 2025-10-17; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Heart Failure - NYHA II - IV
Keywords: Fibroscan; Vibration Control Transient Elastography; Liver Stiffness Measurement; Guided VCTE
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a pivotal, global, prospective, cross-sectional, multicentric clinical investigation
Masking Description: To minimize bias in clinical performance evaluation, the participant and operator of the device under test will be blinded to the clinical reference standard (ie, CVP as assessed by invasive hemodynamic catheter) result.
  The FibroScan operator will not be the same as the hemodynamic catheterization operator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Full Cohort (Experimental): This population will be defined by patients fulfilling all inclusion and exclusion criteria.
  Interventions: Device: FibroScan; Procedure: Right-sided Heart Catheterization; Procedure: Transthoracic echocardiography; Biological: Blood Sample Analysis

INTERVENTIONS:
Device: FibroScan — At Day 0: 1 FibroScan examination to collect Liver Stiffness Measurement (LSM)
Procedure: Right-sided Heart Catheterization — at Day 0: Right-sided Heart Catheterization (RHC) to measure Central Venous Pressure (CVP)
Procedure: Transthoracic echocardiography — at Day 0 assessment of cardiac function
Biological: Blood Sample Analysis — At Day0: To assess baseline organ function that may impact participant safety, and blood samples for clinical laboratory tests

SUMMARY:
This is a pivotal, global, prospective, cross-sectional, multicentric clinical investigation designed to explore a non-invasive, reliable alternative to invasive, catheter-based hemodynamic assessments, which are associated with procedural risks and limited applicability in certain participant populations.

DETAILED DESCRIPTION:
CHF, as defined by the American College of Cardiology and the American Heart Association, is "a complex clinical syndrome that results from any structural or functional impairment of ventricular filling or ejection of blood." These patients will often develop congestion that may require urgent hospitalization, especially if pulmonary congestion is present. However, congestion can be difficult to assess, especially when symptoms are mild, or in patients nearing discharge from an HF hospitalization.8 Increased cardiac filling pressures, including the CVP, often silently precede the appearance of congestive symptoms by days resulting in hepatic congestion.

Invasive methods, such as RHC, remain the gold standard method of measuring CVP, offering accurate and direct hemodynamic data. However, RHC requires specialized training and invasive vascular access and is associated with procedural risks including bleeding, infection, arrhythmia, and patient discomfort.

Echocardiography is the most common non-invasive adjunct tool for estimating CVP and assessing cardiac function. It evaluates indirect parameters, right atrial size, IVC diameter, and collapsibility to detect elevated CVP.

LSM by VCTE™ has emerged as a novel non-invasive approach to detecting elevated CVP indirectly. Liver elastography relies on imaging techniques to assess LSM, with high values equating to increased stiffness. While this was developed to assess fibrosis in chronic liver diseases, LSM also reflects increased CVP and hepatic congestion. Multiple studies have shown promising correlations between increased liver stiffness and invasively measured CVP, indicating a potential clinical strategy for detecting hemodynamic congestion non-invasively.

Given these considerations, the current clinical investigation aims to evaluate the 13.3 kPa cutoff performance of LSM with FibroScan (Echosens, Paris, France) to diagnose elevated CVP (>10 mm Hg).

ELIGIBILITY:
Inclusion Criteria:

1. Have read, understood, and signed the informed consent form (ICF)
2. Be ≥18 years of age at the time of screening
3. Have suspected or diagnosed acute or chronic HF and be scheduled to undergo right-sided cardiac catheterization

Exclusion Criteria:

1. Inability to consent
2. Chronic liver disease (self-reported alcohol use >14 drinks/week in females and >21 drinks/week in males), positive hepatitis C virus serology, positive hepatitis B surface antigen, autoimmune hepatitis, hemochromatosis, or cholestatic disease)
3. BMI >40 kg/m2
4. Fontan-type circulation
5. Ascites
6. Heart transplantation
7. Pregnancy, breastfeeding, or intent to become pregnant during the study
8. Intent to donate/bank or retrieve eggs (ova, oocytes) or donate sperm during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with elevated CVP (>10 mm Hg) who are correctly identified by LSM (cutoff of 13.3 kPa) [Sensitivity] | at Day 0
  Sensitivity (true positive rate) = TP / (TP + FN)
Proportion of individuals without elevated CVP (>10 mm Hg) who are correctly identified by LSM (cutoff of 13.3 kPa) [Specificity] | at Day 0
  Specificity (1 - false negative rate) = TN / (TN + FP)

SECONDARY OUTCOMES:
Proportion of individuals correctly identified by LSM (Youden index) for the diagnosis of elevated CVP (>10 mm Hg) | at Day 0
Proportion of individuals correctly identified by LSM (Youden index) for the diagnosis of abnormal IVC diameter | at Day 0
Logistic regression model to identify clinical, laboratory, and echocardiographic factors associated with LSM/CVP discordance. | at Day 0
Correlation between LSM and echocardiographic parameters evaluated with Pearson or Spearman correlation coefficients | at Day 0
  * Unit of measure: Pearson or Spearman coefficient
  * Measurement tool: linear regression
Correlation between LSM and NT-proBNP evaluated with Pearson or Spearman correlation coefficients | at Day 0
  * Unit of measure: Pearson or Spearman coefficient
  * Measurement tool: linear regression
Correlation between LSM and CA-125 evaluated with Pearson or Spearman correlation coefficients | at Day 0
  * Unit of measure: Pearson or Spearman coefficient
  * Measurement tool: linear regression
Correlation between LSM and clinical parameters evaluated with Pearson or Spearman correlation coefficients | at Day 0
  * Unit of measure: Pearson or Spearman coefficient
  * Measurement tool: linear regression
Proportion of individuals correctly identified for the diagnosis of elevated CVP (>10 mm Hg) compared between LSM, echocardiography parameter and NT-proBNP using DeLong's test for correlated ROC curves | at Day 0

OTHER OUTCOMES:
Number of patient presenting at least one adverse event | 7 days

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Keck Medicine of USC-Norris Healthcare Center - Transplant Clinic, Los Angeles, California
  - University of Minnesota, Minneota, Minnesota
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center - Clinical Heart and Vascular Center - West Campus Building 3 Location, Dallas, Texas
- Centre Hospitalier Universitaire (CHU) de Rennes - Hopital de Pontchaillou, Rennes, Ile Et Vilaine, France
- Deutsches Herzzentrum der Charité (DHZC) - Klinik fuer Herz-, Thorax- und Gefaesschirurgie, Berlin, Germany
- Uniwersytet Medyczny im. Piastow Slaskich we Wroclawiu, Instytut Chorob Serca, Wroclaw, Basse-Silésie, Poland